CLINICAL TRIAL: NCT05510830
Title: A Study of the Value of Diagnostic Cervical Conization for Persistent Infection or Integration of Human Papillomavirus
Brief Title: Diagnostic Cervical Conization for Persistent Infection or Integration of HPV
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Li Shuang, Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TJ-IRB20220769
Record Dates: First submitted 2022-08-16; First posted 2022-08-22 (Actual); Last update posted 2022-09-08 (Actual); Status verified 2022-09

CONDITIONS: Human Papilloma Virus Infection; Human Papilloma Virus Integration; Cervical Intraepithelial Neoplasia; Cervical Cancer; Cervical Conization
Keywords: HPV persistent infection; HPV integration; diagnostic cervical conization
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): The patients who meet the inclusion criteria will receive diagnostic cervical conization for pathological examinations. Then they will be followed up for at least two years with every six months' return to our clinics to test HPV and colposcopy if necessary.
  Interventions: Procedure: diagnostic cervical conization

INTERVENTIONS:
Procedure: diagnostic cervical conization — For the patients who met the inclusion criteria, the gynecologists perform cervical conization and pathological examinations. Then the patients will be followed-up for at least two years with the tests of cervical TCT & HPV, and colposcopy if necessary. The data will be analyzed and see if the patients with high risk factors benefit from the surgery or not.

SUMMARY:
For the patients with cervical persistent infection or integration of HPV, we has designed a program to perform cervical conization for certain patients to earlier and better diagnose and cure the diseases of HPV infection and related cervical intraepithelial neoplasia/cancer.

DETAILED DESCRIPTION:
For the patients with cervical persistent infection or integration of human papillomavirus, the incidence of suffering cervical cancer or percancerous lesions increases. As the biopsy guided by colposcopy might miss some lesions, the cervical conization plays a role for the patients with high risk factors to diagnose the related cervical diseases. In this study, we has designed a program to perform cervical conization for certain patients to earlier and better diagnose and cure the diseases of HPV infection and related cervical intraepithelial neoplasia/cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The patients are referred to colposcopy and biopsy examinations due to abnormal cervical screening results with no precancerous lesions discovered by pathology.
2. The cervical precancerous lesions are highly suspected by clinicians with one or more following risk factors:

   * The course of HPV type 16/18 persistent infection is more than two years.
   * The integration reads of HPV is more than 15.
   * The impression of colposcopy indicates precancerous lesions.
   * The cervical TCT indicates ASC-H/HSIL/SCC/AGC-FN/AIS/AC.

Exclusion Criteria:

1. Pregnant women.
2. Vaginal intraepithelial neoplasia is highly suspected by colposcopy and pathological examinations.
3. The patients are suffering malignant tumors of other system and have not been cured.
4. There is acute inflammation of the lower genital or anal tract.
5. The patients' health will be severely harmed by the colposcopy and cervical conization due to some circumstances such as severe insufficiency of liver and kidney function, blood diseases and acute inflammation of other systems.

Ages: 25 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of discovering concealed cervical cancer or percancerous lesions | up to 2 months after recruited
  The pathological examinations of the cervical conization might discover some concealed cervical cancer or precancerous lesions which could not be discovered by biopsy guided by colposcopy.
The incidence of HPV clearance after the cervical conization | Through the study completion, an average of 3~5 years
  After the cervical conizations, the patients will be arranged for follow-up every six months and HPV will be tested to see if the virus is cleared or not

CONTACTS AND LOCATIONS:
Overall Officials: Shuang Li, M.D, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Every six month, we will check if there is a new subject recruited in the study and update the data.
Supporting Information: Study Protocol, SAP, ICF, CSR